CLINICAL TRIAL: NCT05637034
Title: Clinical Applications of Fibroblast Activation Protein Inhibitor-Based Dimeric Radiotracer 68Ga-DOTA-F2 PET/CT Imaging for Malignant Tumors
Brief Title: 68Ga-DOTA-F2 PET/CT in Patients With Various Types of Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: I-22PJ292
Record Dates: First submitted 2022-11-27; First posted 2022-12-05 (Actual); Last update posted 2022-12-05 (Actual); Status verified 2022-11

CONDITIONS: Tumor, Solid
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 68Ga-DOTA-F2 PET/CT and 18F-FDG (Experimental): Each subject receive a single intravenous injection of 68Ga-DOTA-F2 and 18F-FDG, and undergo PET/CT imaging within the specified time.
  Interventions: Diagnostic Test: 68Ga-DOTA-F2 PET/CT and 18F-FDG

INTERVENTIONS:
Diagnostic Test: 68Ga-DOTA-F2 PET/CT and 18F-FDG — Each subject receive a single intravenous injection of 68Ga-DOTA-F2 and 18F-FDG, and undergo PET/CT imaging within the specified time.

SUMMARY:
To evaluate the potential usefulness of 68Ga-DOTA-F2 positron emission tomography/computed tomography (PET/CT) for the diagnosis of primary and metastatic lesions in various types of cancer, compared with 18F-FDG PET/CT.

DETAILED DESCRIPTION:
Quinoline-based fibroblast activation protein (FAP) inhibitors (FAPIs; e.g., FAPI-04 and FAPI-46), which have shown promising results in the diagnosis of cancer and various other diseases in recent years, have become the focus of much productive research. Despite this, one major issue is that these FAPI molecules have a relatively short tumor retention time, which may limit their use in targeted radionuclide therapy applications. As a result, 68Ga-DOTA-F2, a novel dimeric FAPI molecule, was developed to increase tracer uptake and retention in tumors for potential therapeutic or theranostic applications. In preclinical study, 68Ga-DOTA-F2 has shown better tumor uptake and longer tumor retention time than 68Ga-FAPI in mouse tumor models. Our study will assess image quality and evaluate the diagnostic performance of 68Ga-DOTA-F2. Patients with histologically confirmed malignant tumors will be prospectively recruited in this study.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is aged 18 years or older
2. Signed Informed Consent
3. Subject is pathologically confirmed with a malignant tumor
4. Subject is judged to be in good general condition by the investigator based on medical history, physical examination including vital signs and clinical laboratory tests, besides the diagnosis of malignant tumor
5. Female subjects should be post-menopausal or surgically sterile or using effective contraceptive with the negative pregnancy test

Exclusion Criteria:

1. Subject has a previous or ongoing recurrent or chronic disease, other than malignant tumor, at high risk to interfere with the evaluation of the trial according to the judgment of the investigator
2. Subject with non-malignant lesions;
3. Subject with the inability or unwillingness of the research participant, parent or legal representative to provide written informed consent.
4. Subject is potentially pregnant (serum and urinary hCG test will be performed in women where pregnancy is not excluded) or is breast-feeding

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-09-15 (Actual); Primary Completion 2023-09-15 (Estimated); Study Completion 2023-09-15 (Estimated)

PRIMARY OUTCOMES:
Standardized uptake value (SUV) | through study completion, an average of 1 year
  Standardized uptake value (SUV) of 68Ga-DOTA-F2 and 18F-FDG for each primary tumor of subject or suspected lymph metastasis
Lession detection ability | through study completion, an average of 1 year
  Lession number detected by 68Ga-DOTA-F2 and 18F-FDG PET/CT

SECONDARY OUTCOMES:
Sensitivity | through study completion, an average of 1 year
  The sensitivity of 68Ga-DOTA-F2 PET/CT and 18F-FDG PET/CT
Specificity | through study completion, an average of 1 year
  The specificity of 68Ga-DOTA-F2 PET/CT and 18F-FDG PET/CT
Radiation Dosimetry | 30 days
  Mean absorbed radiation doses were estimated using the source and target organ framework. Five patients with different cancers underwent serial 68Ga-DOTA-F2 PET/CT scans at five-time points following radiotracer injection: 5 minutes, 15 minutes, 30 minutes, 1 hour, and 3 hours. The source organs consisted of the kidneys, bladder, liver, heart, spleen, bone marrow, uterus, and body remainder. OLINDA/EXM software was used to fit and integrate the kinetic organ activity data to yield total body and organ time-integrated activity coefficients/residence times and finally organ absorbed doses.

CONTACTS AND LOCATIONS:
Overall Officials: Fang Li, MD, Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Peking union medical college hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No